CLINICAL TRIAL: NCT03750513
Title: Pilot Trial of LET Optimized IMPT for Pediatric Patients With Ependymoma
Brief Title: LET Optimized IMPT in Treating Pediatric Patients With Ependymoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0344; NCI-2018-02519 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0344 (Other: M D Anderson Cancer Center); P30CA016672 (NIH); U19CA021239 (NIH)
Record Dates: First submitted 2018-11-15; First posted 2018-11-23 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Anaplastic Ependymoma; Ependymoma
MeSH Terms: conditions — Ependymoma | interventions — Linear Energy Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (LET optimized IMPT) (Experimental): Patients receive LET optimized IMPT for up to 6 weeks.
  Interventions: Radiation: Linear Energy Transfer-Optimized Intensity Modulated Proton Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Radiation: Linear Energy Transfer-Optimized Intensity Modulated Proton Therapy — Given LET optimized IMPT
  Other Names: LET-Optimized IMPT; LET-Optimized Intensity Modulated Proton Therapy; Linear Energy Transfer (LET)-Optimized Intensity Modulated Proton Therapy (IMPT)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial studies the side effects of linear energy transfer (LET) optimized image modulated proton therapy (IMPT) in treating pediatric patients with ependymoma. Radiation therapy such as LET optimized IMPT, uses proton beams to kill tumor cells and shrink tumors without damaging surrounding normal tissues.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of linear energy transfer (LET) optimized image modulated proton therapy (IMPT) (bio-IMPT) for pediatric patients with ependymoma.

SECONDARY OBJECTIVES:

I. To utilize advanced multiparametric magnetic resonance (MR) imaging to identify imaging biomarkers of structural and biological changes after proton therapy in pediatric ependymoma patients.

II. To compare quantitative image biomarkers in patients treated with bio-IMPT and standard proton therapy using a voxel level analysis.

III. To test and evaluate the validity of relative biological effectiveness (RBE) models and enhance their precision based on prospectively collected clinical image biomarkers.

IV. To evaluate acute and late toxicities, including pseudoprogression and symptom burden, in patients treated with bio-IMPT.

V. To estimate progression-free survival (PFS) and overall survival (OS). VI. To evaluate disease outcomes following the use of a simultaneous integrated boost (SIB) for pediatric ependymoma patients with gross residual disease following surgery.

OUTLINE:

Patients receive LET optimized IMPT for up to 6 weeks.

After completion of study treatment, patients are followed up at 1 month, then every 3 months for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Previous pathologic confirmation of ependymoma, World Health Organization (WHO) grade II or III
* Disease must be confined to the brain (no evidence of spread on MR imaging of the spine or on staging lumbar puncture)
* Patient may not receive chemotherapy concurrent with radiation
* Signed informed consent by patient and/or parents or legal guardian
* Lansky performance status score of 50 -100

Exclusion Criteria:

* Patients with previous radiation therapy to the brain
* Ependymoma of the spine
* Disseminated ependymoma requiring craniospinal radiation therapy
* Pregnancy
* Inability to undergo MR imaging
* Inability to receive gadolinium-based contrast agent

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 6 months post treatment
  The safety of linear energy transfer-optimized intensity modulated proton therapy will be defined by treatment failures which include imaging changes consistent with necrosis in the presence of Common Terminology Criteria for Adverse Events version 4.03 symptoms of grade 3 brain necrosis and/or local recurrence within the first 6 months from the end of proton therapy.

SECONDARY OUTCOMES:
Identify imaging biomarkers of structural and biological changes after proton therapy | Up to 24 months post-treatment
  Descriptive statistics will be used to summarize the study data.
Quantitative image biomarkers | Up to 24 months post-treatment
  Descriptive statistics will be used to summarize the study data.
Validity of relative biological effectiveness models | Up to 24 months post-treatment
  Descriptive statistics will be used to summarize the study data.
Incidence of late and acute toxicities | Up to 24 months post treatment
  Descriptive statistics will be used to summarize the study data. For each study cohort, we will tabulate treatment- failures and other relevant clinically-related features. Interval estimates for proportions will be provided using exact 95% confidence intervals.
Progression-free survival | Up to 24 months post treatment
  The method of Kaplan and Meier will be used to provide estimates.
Overall survival | Up to 24 months post treatment
  The method of Kaplan and Meier will be used to provide estimates.
Disease outcomes following the use of a simultaneous integrated boost | Up to 24 months post-treatment
  Descriptive statistics will be used to summarize the study data.

CONTACTS AND LOCATIONS:
Overall Officials: David R Grosshans, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org